CLINICAL TRIAL: NCT04156529
Title: The Effect of Two Different Feeding Positions During Tube Feeding on Stress, Pain Level and Feeding Tolerance of Preterm Infants
Brief Title: The Effect of Feeding Positions During Tube Feeding on Stress, Pain Level and Feeding Tolerance of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Serap Ceylan (Other)
Responsible Party: Sponsor-Investigator, Sibel Serap Ceylan, Principal Investigator, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PamukkaleUniversity
Record Dates: First submitted 2019-10-11; First posted 2019-11-07 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Pain; Stress; Enteral Feeding Intolerance
Keywords: body position; enteral feeding intolerance; nursing care; pain; stress
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESU position (Experimental): Firstly, the semi-elevated supine position was given to participants during tube feeding
  Interventions: Behavioral: ESU position; Behavioral: ESRL position
- ESRL position (Experimental): Firstly, the semi-elevated right lateral position was given to participants during tube feeding
  Interventions: Behavioral: ESU position; Behavioral: ESRL position

INTERVENTIONS:
Behavioral: ESU position — Semi-elevated supine (ESU) position was given during tube feeding
Behavioral: ESRL position — Semi-elevated right lateral (ESRL) position was given during tube feeding

SUMMARY:
Premature infants have a need for an orogastric or nasogastric feeding tube because of the immaturity of coordination between suck-swallow and breathing. Tube feeding could cause feeding intolerance and stress. One of the recommendations to prevent feeding intolerance is giving suitable position during tube feeding. Also, feeding intolerance is related to stress. The aim of this study was to investigate the effect of semi-elevated supine (ESU) and semi-elevated right lateral (ESRL) positions on the stress, pain levels and feeding tolerance of premature infants during the tube feeding (TF). This was a clinical trial with a crossover design in which subjects randomly received a sequence of either ESU position or ESRL position, during the TF.

DETAILED DESCRIPTION:
Purpose: The aim of this study was to investigate the effect of semi-elevated supine (ESU) and semi-elevated right lateral (ESRL) positions on the stress, pain levels and feeding tolerance of premature infants during the tube feeding (TF).

Method: This was a clinical trial with a crossover design in which subjects randomly received a sequence of either ESU position or ESRL position, during the TF. The sample size calculation was based on the crossover design. It assumed criteria that included the expectation of minimal differences in the average pain and stress score, 1.0; a difference of 2.0 in the standard deviation between ESU and ESRL positions; power, 0.80 and p < .05. The sample size was calculated to be 34 participants. The inclusion criteria for participants were 30-34 weeks gestational age, stable vital signs, no oral feeding skills, feeding by orogastric tube, and had parental consent. Exclusion criteria were respiratory distress, congenital anomalies, necrotizing enterocolitis history, neurological and cardiological problems, receiving analgesic, sedative, or muscle relaxant medication that may affect pain and stress. The position to be given to the participants during TF first was determined by randomization. The sequence of feeding position was randomized by computer. Sixteen of the infants started TF with ESU position, whereas the other 18 started with ESRL position.

The study data were collected with "Descriptive Properties Form of Premature Newborn", Premature Newborn Follow-up Form", "Newborn Stress Scale", "ALPS-Neo Newborn Pain and Stress Assessment Scale".

For each participant, two feeding positions were applied at consecutive feeding time. Feeding tolerance was assessed by abdominal circumference measurements and checking gastric residuals. The abdominal circumference of the participants was measured with a tape measure before and after TF. Vital signs and oxygen saturation levels were measured before, during and after TF. The stress and pain levels of the participants were evaluated independently by the researchers before, during and after TF. Significance level p <0.05 was used for all statistical analyses. Ethics committee approval, written permission from institutions and families were obtained for conducting the study.

ELIGIBILITY:
Inclusion Criteria:

* 30-34 weeks gestational age,
* stable vital signs,
* no oral feeding skills,
* feeding by orogastric tube,
* had parental consent

Exclusion Criteria:

* respiratory distress,
* congenital anomalies,
* necrotizing enterocolitis history,
* neurological and cardiological problems,
* receiving analgesic, sedative, or muscle relaxant medication that may affect pain and stress

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Neonatal pain | Four month
  ALPS-Neo Newborn Pain and Stress Assessment Scale was used. The ALPS-Neo is a five-item scale including facial expression, breathing pattern, tone of extremities, hand and foot activity, and level of activity. The lowest and the highest scores obtainable from the scale are 0 and 10, respectively. As the score increases, stress and pain increase.
Neonatal stress | Four month
  Newborn Stress Scale was used. The scale includes eight items: face expression, color, respiration, activity level, consolation, muscle tone, extremities, and posture. Each item is scored on the scale 0-2. The minimum score is 0 and the maximum score is 16. As the score increases, the stress level of the infant increases.
Feeding intolerance | Four month
  Abdominal circumference measurements and checking gastric residuals. The abdominal circumference of the participants was measured with a tape measure before and after TF.

SECONDARY OUTCOMES:
Heart Rate | Four month
  A pulse oximetry probe was attached to the foot to measure heart rate. The number of heartbeats per minute was observed from the pulse oximetry monitor.
Oxygen Saturation | Four month
  Oxygen saturation (SpO2) was obtained using a pulse oximetry device. Pulse oximetry measures peripheral arterial oxygen saturation (%) as a surrogate marker for tissue oxygenation.
Respiratory Rate | Four month
  The respiratory rate is the number of breaths a person takes per minute. Respiratory rate was measured by observation.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Serap Ceylan, Study Director — Pamukkale Univesity
Locations (1):
- Sibel Serap Ceylan, Denizli, Turkey (Türkiye)

REFERENCES:
- [Result] Khatony A, Abdi A, Karimi B, Aghaei A, Brojeni HS. The effects of position on gastric residual volume of premature infants in NICU. Ital J Pediatr. 2019 Jan 8;45(1):6. doi: 10.1186/s13052-018-0591-9. PMID 30621733
- [Result] Dsilna A, Christensson K, Gustafsson AS, Lagercrantz H, Alfredsson L. Behavioral stress is affected by the mode of tube feeding in very low birth weight infants. Clin J Pain. 2008 Jun;24(5):447-55. doi: 10.1097/AJP.0b013e3181633fd6. PMID 18496310